CLINICAL TRIAL: NCT01471587
Title: Fibre Specific Signalling in the Locomotor Myopathy of COPD
Brief Title: Fibre Specific Signalling in the Locomotor Myopathy of Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ERICA WP1b
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — muscle and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with COPD

SUMMARY:
Skeletal muscle is composed of two fibre types which are intertwined. Skeletal muscle weakness, particularly of the walking muscles, is an important complication of Chronic Obstructive Pulmonary Disease (COPD) but so far the investigators do not know what mechanisms drive the process.

All existing studies have investigated signalling pathways in the whole muscle so they have been forced to consider type I and type II fibres together. It is possible that disease selectively affects one fibre type, most likely type I fibres which are in fact lost in COPD patients. For this reason mechanisms of disease may have been overlooked by current studies.

The applicants have acquired the technology which allows type I and type II fibres in a muscle specimen to be split (by laser capture microdissection) and so signalling pathways can be assessed separately in type II and type I fibres which is what this proposal sets out to do.

The proposal therefore aims to capture well characterised clinical data from 60 COPD patients and 20 age matched controls, from whom a biopsy of the main walking muscle, the quadriceps, will be taken. In the samples the investigators will assess at a fibre specific level inflammatory signalling. Surplus material will be retained for subsequent fibre specific analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40 - 90 years inclusive.
* A clinical diagnosis of COPD based on spirometry (FEV1/FVC ratio < 70% on entry to the study with FEV1 < 80% predicted)

Exclusion Criteria:

* History or current diagnosis of alpha 1-anti-trypsin deficiency, asthma, lung cancer, bronchiectasis or other significant respiratory disease (including treated TB in the past 10 years)
* Contraindication to biopsy for research purpose (e.g. use of anticoagulant in the 1 week prior to biopsy)
* Joint or neurological disease which on its own would preclude exercise

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COPD
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
inflammatory signalling at a fibre specific level | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Polkey, PhD FRCP, Principal Investigator — RBHFT
Locations (1):
- Royal Brompton Hospital, London, UK, United Kingdom

REFERENCES:
- [Derived] Buttery SC, Mohan D, Fisk M, Hopkinson NS, Tal-Singer R, Wilkinson IB, Polkey MI. Longitudinal follow-up of quadriceps strength and function in a COPD cohort after 3 years. Eur Respir J. 2017 Aug 10;50(2):1700707. doi: 10.1183/13993003.00707-2017. Print 2017 Aug. No abstract available. PMID 28798091